CLINICAL TRIAL: NCT06769906
Title: Effectiveness of Individualized Automatic Target Coaching Message Based on the Metrics of Continuous Glucose Monitoring and Depressive Symptom in Patients With Insulin-treated Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Effectiveness of Individualized Automatic Coaching Message for Glycemic Management and Depressive Symptom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gyuri Kim, Principal Investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SamsungMC_ENDO_3
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Type 2; Continuous Glucose Measurement; Depressive Symptom
Keywords: Behavioral Symptom; Glucose Metabolism Disorders; Endocrine System Diseases; Diabetes Mellitus, Type 2; Continuous glucose monitoring; Depression; Diabetes Mellitus; Metabolic Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Behavioral Symptoms; Glucose Metabolism Disorders; Endocrine System Diseases; Diabetes Mellitus; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized automatic coaching message for glycemic management and depressive symptoms (Experimental): The study will enroll insulin-treated patients with type 2 diabetes who are already receiving standard care and diabetes management through outpatient visits. For 12 weeks, the intervention group and control will apply continuous glucose monitoring. The intervention group will receive weekly personalized coaching messages for glycemic management based on data from continuous glucose monitoring and bi-weekly personalized coaching messages for depressive symptoms based on depression questionnaires for 12 weeks.
  Interventions: Other: Individualized automatic coaching message for glycemic management and depressive symptom
- Control (No Intervention): The control group will continue their existing treatment and wear a continuous glucose monitoring device, responding to both surveys by accessing the survey link sent to their cell phone. This will allow for the assessment of baseline satisfaction (DTSQ) and depressive symptoms (PHQ-9).

INTERVENTIONS:
Other: Individualized automatic coaching message for glycemic management and depressive symptom — For 12 weeks, the intervention group will apply continuous glucose monitoring system and receive weekly personalized coaching messages for glycemic management based on data from continuous glucose monitoring and bi-weekly personalized coaching messages for depression symptoms based on depression questionnaires.
  Arms: Individualized automatic coaching message for glycemic management and depressive symptoms

SUMMARY:
This is a 12-week, single-center, randomized, prospective, confirmatory study of effectiveness of the individualized automatic coaching messages for glycemic management based on continuous glucose monitoring and depressive symptom in insulin-treated patients with type 2 diabetes.

DETAILED DESCRIPTION:
This study will enroll patients with type 2 diabetes who are insulin-treated outpatient care at the Department of Endocrinology and Metabolism, Samsung Medical Center. For 12 weeks, both intervention and control groups will apply continuous glucose monitoring system. The intervention group will receive weekly personalized coaching messages for glycemic management based on data from continuous glucose monitoring and bi-weekly personalized coaching messages for depressive symptoms based on depression questionnaires. The control group will not receive the coaching messages. The aim of this study is to evaluate whether the efficacy of individualized automatic target coaching messages based on continuous glucose monitoring metrics and depressive symptom assessments is superior to those who do not receive the messages in insulin-treated patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the use of a continuous glucose monitor has been determined based on the medical judgment of the attending physician.
* Insulin-treated type 2 diabetes patients, age 18-80 years old.
* Patients who have not changed their diabetes medication in the past 2 months.
* Patients with a glycated hemoglobin level between 6.5% and 12.0% within the last 3 months.
* Patients currently receiving insulin injection therapy, including basal insulin.
* Patients who have access to KakaoTalk via smartphone and are able to communicate with it.
* Voluntarily agreed to participate in this clinical study.

Exclusion Criteria:

* Steroid and immunosuppressant users. But it can be included if patients continuously maintain same drug dose at least three months.
* Patients who are currently taking weight control medications.
* Breastfeeding or pregnant patients
* Patients who do not voluntarily consent to the study
* Anyone deemed unsuitable by the investigator to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Time In Range | Week 12
  Derived from continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Diabetes treatment satisfaction | Week 12
  Diabetes Treatment Satisfaction Questionnaire (DTSQ);
  Minimum and Maximum Values: The DTSQ consists of eight items, with six items measuring satisfaction scored on a 0-6 scale (where 0 is very dissatisfied and 6 is very satisfied). The scores for these six items are summed, giving a total score range from 0 to 36.
  Higher Scores: Higher scores on the DTSQ indicate better satisfaction with diabetes treatment. A higher total score suggests greater satisfaction, while a lower score indicates dissatisfaction.
Depressive symptoms | Week 12
  Patient Health Questionnaire-9 (PHQ-9); Minimum and Maximum Values: The PHQ-9 consists of nine items, each scored from 0 (not at all) to 3 (nearly every day). The scores for each item are summed to give a total score, resulting in a range from 0 to 27.
  Higher Scores: Higher scores on the PHQ-9 indicate worse outcomes, meaning greater severity of depressive symptoms. Lower scores suggest fewer symptoms of depression or none at all.
  Interpretation of Scores:
  0-4: Minimal or no depression; 5-9: Mild depression; 10-19: Moderate depression; 20-27: Severe depression
Time In Tight Range | Week 12
  Derived from CGM
Level of glycated Hemoglobin | Week 12
  Derived from blood measurement
Time Above Range | Week 12
  Derived from CGM
Time Below Range | Week 12
  Derived from CGM
Coefficient of Variation | Week 12
  Derived from CGM
Glycemic Management Indicator | Week 12
  Derived from CGM

OTHER OUTCOMES:
Level of Albuminuria | Week 12
  Urine creatinine-to-albumin ratio
Level of Glycated albumin | Week 12
  Glycated albumin
Level of triglycerides | Week 12
  Level of triglycerides from blood measurement
Level of total cholesterol | Week 12
  Level of total cholesterol from blood measurement
Level of HDL (high density lipoprotein) cholesterol | Week 12
  Level of HDL cholesterol from blood measurement
Level of LDL (low density lipoprotein) cholesterol | Week 12
  Level of LDL cholesterol from blood measurement

CONTACTS AND LOCATIONS:
Overall Officials: GYURI KIM, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No